CLINICAL TRIAL: NCT04773873
Title: Randomized Controlled Clinical Trial (RCT) of Implant-retained Monolithic Chairside-made CAD-CAM Hybrid Abutment Single Crowns
Brief Title: Implant Retained CAD-CAM Ceramic Crowns
Acronym: RCT-Scherrer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Scherrer (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Sponsor-Investigator, Susanne Scherrer, Associate Professor, Head of Biomaterials, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-Hybrid abutment
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: 90 RCT crowns will be allocated in three groups of ceramic materials (3 materials) and at two tooth locations (premolar and molar)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Porcelain fused to metal (PFM) (Active Comparator): Implant screw-retained PFM crown fabricated by a laboratory using a gold coping cast-on synOcta gold abutment (Ceramicor) for wide (WN) or regular (RN) neck
  Interventions: Device: PFM Crowns on gold coping cast-on
- Arm 2: Hybrid abutment Lithium disilicate (e.max CAD) (Experimental): Hybrid crown abutment: chairside-made perforated CAD-CAM Lithium disilicate crown (IPS e.max CAD LT A16) adhesively cemented to a TiBase and screw-retained to a Straumann titanium implant (regular and wide neck)
  Interventions: Device: hybrid abutment lithium disilicate crown
- Arm 3:Hybrid abutment ceramic polymer infiltrated (Enamic) (Experimental): Hybrid crown abutment: chairside-made perforated CAD-CAM ceramic-polymer infiltrated crown (Enamic) adhesively cemented to a TiBase and screw-retained to a Straumann titanium implant (regular and wide neck)
  Interventions: Device: hybrid abutment ceramic polymer infiltrated crown

INTERVENTIONS:
Device: PFM Crowns on gold coping cast-on — Classic impressions are taken by the operators and sent to one and same laboratory who will deliver all the screw-retained PFM restorations. The crowns will be made using a gold coping cast-on synOcta gold abutment (Ceramicor) for wide (WN) or regular (RN) neck
  Other Names: SynOcta gold coping cast-on (Ceramicor)
  Arms: Arm 1: Porcelain fused to metal (PFM)
Device: hybrid abutment lithium disilicate crown — Intraoral digital impression with respective scanbodies (Sirona) for Cerec OmniCam or Cerec Bluecam over the chosen TiBase. Cerec CAD designing (operator) and CAM milling (Cerec MCXL) of single crowns with perforated blocs (e.max CAD). crystallization/ characterization/ glaze firing for the e.max CAD crown using an oven with specific firing programmes for e.max CAD. Adhesive cementation steps of the ceramic crown onto the TiBase
  Other Names: hybrid abutment e.max CAD
  Arms: Arm 2: Hybrid abutment Lithium disilicate (e.max CAD)
Device: hybrid abutment ceramic polymer infiltrated crown — Intraoral digital impression with respective scanbodies (Sirona) for Cerec OmniCam or Cerec Bluecam over the chosen TiBase. Cerec CAD designing (operator) and CAM milling (Cerec MCXL) of single crowns with perforated blocs (Enamic). Surface polishing with rubber polishers. Adhesive cementation steps of the ceramic crown onto the TiBase
  Other Names: hybrid abutment Enamic
  Arms: Arm 3:Hybrid abutment ceramic polymer infiltrated (Enamic)

SUMMARY:
Newly available ceramic CAD-CAM blocs containing a screw channel for chairside-made crowns to be adhesively cemented to a TiBase abutment and screw-retained to an implant are appealing to the clinician, considering the time efficiency (one appointment) and overall lower costs as no dental laboratory is involved. The hypotheses are that the biological (BOP, PD, PCR, implant bone level) and mechanical outcomes (fracture, loss of retention, wear) are equivalent to implant screw-retained Porcelain-Fused-to-Metal (PFM) crowns over a 5 year observation time.This RCT will provide key information as to the cost/benefit, suitability and/or limitations of these chair-side hybrid-abutment crowns in the posterior region.

DETAILED DESCRIPTION:
This RCT involves the University of Geneva Dental School and four private practices for which the Geneva Hospital Ethic Committee's approval is required. Patients in need for replacement of single unit posterior teeth will be recruited at the Dental School as well as in the 5 private practices based on specific selection criteria. Patients will be randomly assigned to a restorative group using a computer-generated random number table for allocation.

The CAD-CAM blocs containing a screw channel for implant-retained chairside-made single-unit hybrid-abutment crowns are 1) Lithium-disilicate glass-ceramic (e.max CAD) (G1) and 2) feldspath-ceramic infiltrated by polymer (Enamic) (G2). The CAD-CAM crowns are adhesively cemented to titanium base abutments (Ti-base) and screw-retained to Titanium implants (Straumann Standard Plus) in the premolar (RN) and molar region (WN). Controls are screw-retained PFM crowns (G3). The number of crowns in each group is N=30 (15 molars and 15 premolars) which gives a total of 90 crowns for this study.

Participants are recalled after 1 week-10 days after crown insertion (baseline, T0) and then yearly during 5 years (T1-T5). Digital X-Rays are taken at T0, T1, T3 and T5 with repositionable individual resin bite registrations.

ELIGIBILITY:
Inclusion Criteria:

* Absence of relevant medical condition
* Need for a single crown on implant in the molar or premolar region with existing adjacent and antagonist teeth
* No active periodontal or pulpal diseases
* Teeth with good restorations
* Straumann regular (premolar) and wide neck (molar) implants, osseo-integrated for a minimum of 2 months and facial keratinized mucosa width of at least 2 mm
* Patient agrees to return for follow-up examinations during 5 years
* Patient agrees to immediately inform the operator in case of problem

Exclusion Criteria:

* evidence of bruxism
* 2 adjacent implants
* implants placed of-axis

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
survival | 5 years
  The primary aim is to monitor and compare the survival of the two CAD-CAM hybrid abutment crown materials with that of PFM implant screw-retained crowns in the posterior region over a period of 5 years. The survival data is subdivided into "absolute failures" needing replacement of the restoration and "relative failures" which include complications that could be repaired.

SECONDARY OUTCOMES:
Occlusal surface wear | 5 years
  Surface wear generated at occlusal contacts from antagonist teeth will be monitored using silicone replicas of the crowns poured with epoxy resin and gold-cotaed for scanning electron microscopy. The contact wear surface will be expressed in mm^2. The average roughness in Ra values.

OTHER OUTCOMES:
Bone level | T1, T3 and T5 years
  Bone level changes in mm will be monitored through standardized X Rays from registration bites at various time frames (T1, T3 and T5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne S Scherrer, Prof, Dr, Principal Investigator — University of Geneva
Locations (1):
- University Clinics of Dental Medicine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided